CLINICAL TRIAL: NCT01367847
Title: Technology Enhanced Delivery of Treatment for Early Conduct Problems
Brief Title: Technology-Enhanced Helping the Noncompliant Child
Acronym: TE-HNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0740; 1R34MH082956-01A2 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-07 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Child Externalizing Behavior
Keywords: Parenting; Parent-Child Relations; Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Helping the Noncompliant Child (HNC) (Active Comparator): Standard HNC (see HNC Arm/Title) Program plus Technology-Enhancement (smartphones, which are being used for mid-week video calls to check-in re: skill-building, videotaping of family practice of skills at home, daily surveys re: skills practice & child behavior, reminders re: practice & sessions.
  Interventions: Behavioral: Helping the Noncompliant Child (HNC)
- Technology-Enhanced HNC (TE-HNC) (Experimental): Standard HNC (see HNC Arm/Title) Program plus Technology-Enhancement (smartphones, which are being used for mid-week video calls to check-in re: skill-building, videotaping of family practice of skills at home, daily surveys re: skills practice & child behavior, reminders re: practice & sessions.
  Interventions: Behavioral: Technology-Enhanced Helping the Noncompliant Child (TE-HNC)

INTERVENTIONS:
Behavioral: Helping the Noncompliant Child (HNC) — Well-established behavioral parent training program (McMahon & Forehand) for parents of 3 to 8 y.o. children with externalizing problems
  Other Names: HNC
  Arms: Helping the Noncompliant Child (HNC)
Behavioral: Technology-Enhanced Helping the Noncompliant Child (TE-HNC) — Standard HNC program plus technology-enhancements (see description under Arm)
  Other Names: TE-HNC
  Arms: Technology-Enhanced HNC (TE-HNC)

SUMMARY:
This study aimed to examine if technology could enhance the treatment engagement and outcomes of low income parents of 3 to 8 children with externalizing problems.

DETAILED DESCRIPTION:
The aim of this pilot study is to determine whether a technology-enhanced version of an established behavioral treatment protocol, Helping the Noncompliant Child (HNC; McMahon & Forehand), enhances the engagement and treatment outcomes of lower income parents of 3 to 8 children with externalizing problems in treatment. It is predicted that families in both the HNC and technology-enhanced HNC (TE-HNC) programs will evidence significant improvement in parenting behavior and child externalizing problems; however, it is predicted that parent-child dyads in the TE-HNC program will require fewer sessions, will be more likely to be retained in the program, will be more likely to remain engaged in the program (e.g., practicing skills between sessions etc.), and will be more likely to have active involvement from their coparenting partners (i.e., other adults and family members who participate in childrearing).In turn, it is expected that the TE-HNC program will boost treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Lower income
* caregiver/parent is legal guardian
* 3 to 8 year old child
* child meets criteria for externalizing disorder or significant externalizing symptoms

Exclusion Criteria:

* Prior report of child abuse or neglect
* current substance abuse/dependence
* legal guardian reading level less than 8th grade
* child has developmental disability that precludes caregiver utilizing the skills

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Jones, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Jones DJ, Forehand R, McKee LG, Cuellar J, Kincaid C. Behavioral Parent Training: Is There an "App" for That? Behav Ther (N Y N Y). 2010 Apr;33(4):72-77. No abstract available. PMID 22199418
- [Background] Jones DJ, Forehand R, Cuellar J, Kincaid C, Parent J, Fenton N, Goodrum N. Harnessing innovative technologies to advance children's mental health: behavioral parent training as an example. Clin Psychol Rev. 2013 Mar;33(2):241-52. doi: 10.1016/j.cpr.2012.11.003. Epub 2012 Dec 4. PMID 23313761
- [Background] Forehand R, Jones DJ, Parent J. Behavioral parenting interventions for child disruptive behaviors and anxiety: what's different and what's the same. Clin Psychol Rev. 2013 Feb;33(1):133-45. doi: 10.1016/j.cpr.2012.10.010. Epub 2012 Nov 6. PMID 23178234
- [Background] Jones DJ. Future directions in the design, development, and investigation of technology as a service delivery vehicle. J Clin Child Adolesc Psychol. 2014;43(1):128-42. doi: 10.1080/15374416.2013.859082. PMID 24400723
- [Result] Jones DJ, Forehand R, Cuellar J, Parent J, Honeycutt A, Khavjou O, Gonzalez M, Anton M, Newey GA. Technology-enhanced program for child disruptive behavior disorders: development and pilot randomized control trial. J Clin Child Adolesc Psychol. 2014;43(1):88-101. doi: 10.1080/15374416.2013.822308. Epub 2013 Aug 7. PMID 23924046
- [Derived] Loiselle R, Parent J, Georgeson AR, Thissen D, Jones DJ, Forehand R. Validation of the Multidimensional Assessment of Parenting: An application of item response theory. Psychol Assess. 2021 Sep;33(9):803-815. doi: 10.1037/pas0001019. Epub 2021 Apr 26. PMID 33900099
- [Derived] Jones DJ, Loiselle R, Zachary C, Georgeson AR, Highlander A, Turner P, Youngstrom JK, Khavjou O, Anton MT, Gonzalez M, Bresland NL, Forehand R. Optimizing Engagement in Behavioral Parent Training: Progress Toward a Technology-Enhanced Treatment Model. Behav Ther. 2021 Mar;52(2):508-521. doi: 10.1016/j.beth.2020.07.001. Epub 2020 Jul 15. PMID 33622517
- [Derived] Zachary C, Jones DJ, McKee LG, Baucom DH, Forehand RL. The Role of Emotion Regulation and Socialization in Behavioral Parent Training: A Proof-of-Concept Study. Behav Modif. 2019 Jan;43(1):3-25. doi: 10.1177/0145445517735492. Epub 2017 Oct 13. PMID 29029562
- [Derived] Anton MT, Jones DJ, Youngstrom EA. Socioeconomic status, parenting, and externalizing problems in African American single-mother homes: A person-oriented approach. J Fam Psychol. 2015 Jun;29(3):405-415. doi: 10.1037/fam0000086. PMID 26053349
- [Derived] Parent J, Jones DJ, Forehand R, Cuellar J, Shoulberg EK. The role of coparents in African American single-mother families: the indirect effect of coparent identity on youth psychosocial adjustment. J Fam Psychol. 2013 Apr;27(2):252-62. doi: 10.1037/a0031477. Epub 2013 Feb 11. PMID 23398615

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children are participants (i.e., N = # children); however, parents participate with young children in BPT (i.e., reference to parent-child dyads throughout). 22 parent-child dyads enrolled, 3 assigned as practice cases, given the pilot nature of the study (i.e., 19 for analyses), & 4 drop-outs, yielded N = 15 for analysis.
Groups:
- Helping the Noncompliant Child: Helping the Noncompliant Child (HNC) is a well-established behavioral parent training (BPTP program for parents of 3 to 8 year old children with externalizing problems. Children are the target of treatment; however, parents are the mechanism of change. Therefore, parent-child dyads participate.
- TE-HNC: Standard HNC (see HNC Arm/Title) Program plus Technology-Enhancement (smartphones, which are being used for mid-week video calls to check-in re: skill-building, videotaping of family practice of skills at home, daily surveys re: skills practice & child behavior, reminders re: practice & sessions.
Period: Overall Study
Arm/Group | Helping the Noncompliant Child | TE-HNC
Started | 10 | 9
Completed | 8 | 7
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: 22 families enrolled, 3 were therapist practice cases (i.e., 19 remaining for analyses),and 4 were drop-outs, yielding a pilot analysis sample of N = 15
Groups:
- Total: Total of all reporting groups
Arm/Group | Helping the Noncompliant Child | TE-HNC | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.75 (2.12) | 5.57 (1.27) | 5.67 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Minority (Racial and/or Ethnic) | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Retention assesses whether or not the family completed the full treatment program.
Time Frame: Baseline to Post-Intervention (average 8 to 12 weeks)
Population: Given that these analyses focus on retention, the analysis sample is the 19 enrolled parent-child dyads (i.e., including the drop-outs)
Measure: Count of Participants; unit: Participants
Arm/Group | Helping the Noncompliant Child | TE-HNC
Number analyzed (Participants) | 10 | 9
Participants | 8 | 7

2. Primary Outcome: Mean % Sessions Attended as Scheduled
Description: Participation in each weekly session as scheduled was recorded for each family. Mean attendance of scheduled sessions was computed for each parent-child dyad and then for each group. For example, if a parent-child dyad required 8 sessions to master the program skills and attended all 8 sessions as scheduled they would have 100%. If instead, another parent-child dyad also required 8 sessions to complete the program, but half of those were rescheduled at least once. Then the overall average attendance is calculated across the parent-child dyads in each group. Greater scheduled attendance = optimal outcome.
Time Frame: Baseline to Post-Intervention (average 8 to 12 weeks)
Population: Given the pilot nature of study and smalll sample size, intent to treat analyses were not conducted. Rather, analyses were conducted on those parent-child dyads who completed all sessions within each group.
Measure: Mean (Standard Deviation); unit: percentage of scheduled sessions
Groups:
- Helping the Noncompliant Child: Helping the Noncompliant Child (HNC) is a well-established behavioral parent training (BPT) program for parents of 3 to 8 year old children with externalizing problems. Children are the target of treatment; however, parents are the mechanism of change. Therefore, parent-child dyads participate.
Arm/Group | Helping the Noncompliant Child | TE-HNC
Number analyzed (Participants) | 8 | 7
percentage of scheduled sessions | 90 (11) | 97 (5)

3. Secondary Outcome: Mean Post-treatment Score Eyberg Child Behavior Inventory (ECBI)
Description: The ECBI is a 36 item measure frequently used in treatment outcome research with young children, as it it reflects problem behavior in this age range and is sensitive to change. Parents rate the frequency of each problem behavior as occurring 0 = never to 7 = always. Scores can range from 0 to 252 with higher scores reflecting greater problem behaviors.
Time Frame: Baseline to Post-Intervention (average 8 to 12 weeks)
Population: N = 15 parent-child dyads who completed the treatment program.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Helping the Noncompliant Child | TE-HNC
Number analyzed (Participants) | 8 | 7
units on a scale | 91.63 (21.25) | 83.00 (15.34)

4. Secondary Outcome: Mean Sessions for Complete Treatment
Description: Mean number of sessions that parent-child dyads in each group required to master the program skills and complete treatment (Fewer sessions to complete treatment considered more cost-effective as parent-child dyads learning skills more efficiently).
Time Frame: Baseline to Post-Intervention (Average 8 to 12 weeks)
Population: N = 15 parent-child dyads who completed the treatment program.
Measure: Mean (Full Range); unit: Sessions
Arm/Group | Helping the Noncompliant Child | TE-HNC
Number analyzed (Participants) | 8 | 7
Sessions | 10 [7 to 12] | 8 [7 to 10]

5. Secondary Outcome: Mean Consumer Satisfaction
Description: Average parent-reported satisfaction with the treatment program on a project-developed consumer satisfaction scale (Possible range = 11 -77; Higher score = greater satisfaction).
Time Frame: Post-Intervention (Average 8 to 12 weeks)
Population: N = 15 parent-child dyads who completed the treatment program.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Helping the Noncompliant Child | TE-HNC
Number analyzed (Participants) | 8 | 7
score on a scale | 56.56 (2.47) | 59.83 (1.94)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Helping the Noncompliant Child: Helping the Noncompliant Child (McMahon & Forehand), a well-established behavioral parent training program for parents of 3 to 8 year old children with externalizing problems
  Helping the Noncompliant Child (HNC): Well-established behavioral parent training program (McMahon & Forehand) for parents of 3 to 8 y.o. children with externalizing problems
- TE-HNC: Standard HNC Program plus Technology-Enhancement (smartphones, which are being used for mid-week video calls to check-in re: skill-building, videotaping of family practice of skills at home, daily surveys re: skills practice & child behavior, reminders re: practice & sessions.
  Technology-Enhanced Helping the Noncompliant Child (TE-HNC): Standard HNC program plus technology-enhancements (see description under Arm)
Arm/Group | Helping the Noncompliant Child | TE-HNC
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
This is a preliminary randomized control trial with a small sample size and limited statistical power and, thus, findings should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No